CLINICAL TRIAL: NCT01124968
Title: Before and After Study to Assess the Impact of the Use of Virtual Consultation on Frequency of Patient Attendance, and Satisfaction of Patients and Professionals
Brief Title: eConculta: Impact of Virtual Visits in Primary Care
Acronym: eConsulta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Catala de Salut (Other Government)
Responsible Party: Josep Casajuana Brunet (Primary Care Ambit Manager, Barcelona City), Institut Català de la Salut
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: eConsulta
Record Dates: First submitted 2010-05-11; First posted 2010-05-18 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2011-01

CONDITIONS: Adult
Keywords: User-Computer Interface; Office Visits; Primary Health Care; Patient Satisfaction; Job Satisfaction; Health Services Research
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- eConsulta (Experimental): Those patients who are offered to use the eConsulta, a web where they can virtually consult with their primary care doctor or nurse.
  Interventions: Other: eConsulta

INTERVENTIONS:
Other: eConsulta — It is a web specifically designed for the project where elected patients can consult virtually with their primary care physician and within 48 hours have an answer.

SUMMARY:
eConsulta is a before and after quasi-experimental study without control group and its purpose is to asses the impact of virtual visits in primary care on the frequency of attendance of the patients to the primary care centre. The use of virtual consultations should lower the number of face to face visits to primary care. It also should create satisfaction to both users: primary care professionals and patients.

DETAILED DESCRIPTION:
Excess on primary care face to face demands generates a work overload for the professionals, and it could lead to a lower quality of care and less job satisfaction. Not all primary care demands need a face to face encounter so incorporating new technologies into daily practice care such as communication doctor/nurse-patient through a website could be part of the solution. So we designed a study in order to assess the impact of the use of virtual consultation on frequency of attendance and the satisfaction of patients and professionals with the service.

It is a before after quasi-experimental multi-centre study with no control group. Agreed voluntarily to participate 13 primary care centres, 20 primary care physicians, 17 nurses them having 16.720 reference adult patients. We designed a website where participants can access the internet and consult their doctor/nurse, who will answer within 48 hours at maximum. The intervention will last 6 months.

We believe that the site can be useful by both patient and professional. For some types of patient, the use of the site may increase its accessibility, reduce face to face consultations and improve satisfaction, while the professional makes a more efficient practice.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or over
* having a primary care centre assigned
* to have both physician and nurse participating in the project
* to use the same electronic clinical recording software

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16720 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of primary care face to face visits of the patients during the 6 month intervention, compared to the number of face to face visits of the same patient, in a 6 month previous period. | Visits done from 01/06/2010 to 01/12/2010 compared to the himself the same period 1 or 2 years before (depending on the flu)
  Number of face to face visits of each patient (who used the eConsulta web site) to primary care physician or nurse during the 6 months of the intervention (from 01/06/2010 to 01/12/2010) compared to the number of visits of the same patients the same period 1 or 2 years before, depending on the appearance of a swine flu outbreak (2009 if there is a swine flu outbreak or 2008 if there is not). The information source of the number of visits will be the electronic clinical record, which is the same in all the practices participating.

SECONDARY OUTCOMES:
Measure the doctor/nurse satisfaction | At the end of the study, 01/12/2010
  Satisfaction with the whole service with a 10 point scale. Items:
  1. Are you satisfied with the eConsulta?
  2. It is easy to use the web?
  3. Has it been easy to integrate it with the daily practice?
Measure the patient satisfaction | At the end of the study, 01/12/2010
  Satisfaction with the whole service with a 10 point scale. Items:
  1. Are you satisfied with the eConsulta?
  2. It is easy to use the web?
  3. Would you use it in the future?

CONTACTS AND LOCATIONS:
Overall Officials: Josep Casajuana, Principal Investigator — Institut Català de la Salut; Maria A Casas, Study Chair — Institut Català de la Salut; Rosa Chumillas, Study Chair — Institut Català de la Salut; Mireia Fàbregas, Study Chair — Institut Català de la Salut; Ana I Garaikoetxea, Study Chair — Institut Català de la Salut; Maria I Garrido, Study Chair — Institut Català de la Salut; Yolanda Lejardi, Study Chair — Institut Català de la Salut; María J Martínez, Study Chair — Institut Català de la Salut; Maria C Piorno, Study Chair — Institut Català de la Salut; Joan Camús, Study Chair — Institut Català de la Salut
Locations (13):
- Spain (13):
  - EAP Gòtic, Barcelona, Barcelona
  - EAP Ramón Turró, Barcelona, Barcelona
  - EAP El Clot, Barcelona, Barcelona
  - EAP Sant Martí, Barcelona, Barcelona
  - EAP La Sagrera, Barcelona, Barcelona
  - EAP Montnegre, Barcelona, Barcelona
  - EAP Sant Andreu, Barcelona, Barcelona
  - EAP El Carmel, Barcelona, Barcelona
  - EAP Horta, Barcelona, Barcelona
  - EAP Pare Claret, Barcelona, Barcelona
  - EAP Dr. Carles Ribas, Barcelona, Barcelona
  - EAP Congrés, Barcelona, Barcelona
  - EAP Guinardó Baix, Barcelona, Barcelona

REFERENCES:
- [Background] Spielberg AR. On call and online: sociohistorical, legal, and ethical implications of e-mail for the patient-physician relationship. JAMA. 1998 Oct 21;280(15):1353-9. doi: 10.1001/jama.280.15.1353. PMID 9794317
- [Background] Weiss N. E-mail consultation: clinical, financial, legal, and ethical implications. Surg Neurol. 2004 May;61(5):455-9; discussion 459. doi: 10.1016/j.surneu.2003.09.029. PMID 15120220
- [Background] Leong SL, Gingrich D, Lewis PR, Mauger DT, George JH. Enhancing doctor-patient communication using email: a pilot study. J Am Board Fam Pract. 2005 May-Jun;18(3):180-8. doi: 10.3122/jabfm.18.3.180. PMID 15879565
- [Background] Messikomer CM. "Our options have changed. .. we will not call you back". Communicating with my primary care physician. Perspect Biol Med. 2007 Summer;50(3):435-43. doi: 10.1353/pbm.2007.0035. PMID 17660636
- [Background] Roter DL, Larson S, Sands DZ, Ford DE, Houston T. Can e-mail messages between patients and physicians be patient-centered? Health Commun. 2008;23(1):80-6. doi: 10.1080/10410230701807295. PMID 18443995
- [Background] Kjaer NK, Jepsen KL, Ruwald S, Jepsen NP, Nielsen HH. [E-mail communication in general practice]. Ugeskr Laeger. 2005 Nov 21;167(47):4461-5. Danish. PMID 16305766
- [Background] Kuszler PC. A question of duty: common law legal issues resulting from physician response to unsolicited patient email inquiries. J Med Internet Res. 2000 Jul-Sep;2(3):E17. doi: 10.2196/jmir.2.3.e17. No abstract available. PMID 11720940
- [Background] Bovi AM; Council on Ethical and Judicial Affairs of the American Medical Association. Ethical guidelines for use of electronic mail between patients and physicians. Am J Bioeth. 2003 Summer;3(3):W-IF2. doi: 10.1162/152651603322874771. PMID 14735881
- See also: eConsulta — https://econsulta.ics.gencat.cat/public/login/index/ID/